CLINICAL TRIAL: NCT02705170
Title: Index of Microcirculatory Resistance (IMR) Assessment in Patients With New Diagnosis of Left Ventricular Dilatation Without Significant Coronary Artery Lesions: IMPAIRED Pilot Trial
Brief Title: IMR Assessment in Patients With New Diagnosis of Left Ventricle Dilatation
Acronym: IMPAIRED
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Assistant Professor, Interventional Cardiologist, University Hospital of Ferrara
Other Study IDs: 260480
Record Dates: First submitted 2016-03-05; First posted 2016-03-10 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Cardiomyopathies; Microcirculation; Microvessels
Keywords: index of microvascular resistance
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- left ventricle dilatation: The subjects of the investigation will be patients with recent diagnosis of unknown left ventricle dilatation. These subjects received coronary artery angiography as exam suggested by guidelines to discriminate the cause of left ventricle dilatation. In subjects without documentation of coronary artery lesions, the Authors will assess the index of microvascular resistance.
  Interventions: Procedure: index of microvascular resistance

INTERVENTIONS:
Procedure: index of microvascular resistance — Measurement of the index of microvascular resistance in the left anterior descending artery

SUMMARY:
To establish if, in patients with new diagnosis of left ventricular dilatation without documentation at the coronary artery angiography of significant coronary artery lesions, there is a damage of the coronary microcirculation at the IMR (index of microcirculatory resistance) assessment

DETAILED DESCRIPTION:
The Authors will enroll at the moment of coronary artery angiography patients without history of ischemic heart disease and new diagnosis (at transthoracic echocardiography) of left ventricular dilation.

All patients will undergo coronary artery angiography. To be enrolled, it is necessary to have the absence of significant coronary artery stenosis (angiographic evaluation of the lesion >40%) in all the vessels (main and side branch).

The Authors will proceed to perform the evaluation of the index of microvascular resistance (IMR). The target vessel will be the left anterior descending artery.

An intracoronary pressure/temperature sensor-tipped guidewire will be used. Thermodilution curves will be obtained during maximal hyperemia. The IMR will be calculated from the ratio of the mean distal coronary pressure at maximal hyperemia to the inverse of mean hyperemic transit time.

ELIGIBILITY:
Inclusion Criteria:

* new diagnosis of left ventricular dilation (dilatative cardiopathy)
* absence of significant (>40%) coronary artery disease at coronary artery angiography

Exclusion Criteria:

* history of ischemic heart disease
* history of significant valvular disease
* contraindication to hyperemic agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary artery angiography for new diagnosis of left ventricular dilatation (dilatative cardiomyopathy)
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Index of microcirculatory resistance | during coronary artery angiography
  Measurement of IMR in the left anterior descending artery of patients with new diagnosis of left ventricular dilatation and no significant stenosis in epicardial coronary arteries

SECONDARY OUTCOMES:
cardiac death | 1-year
  occurrence of cardiac death at 1 year

OTHER OUTCOMES:
all-cause death | 1-year
  occurrence of all-cause death at 1 year
heart failure | 1-year
  occurrence of hospital admission for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Campo, MD, Principal Investigator — Azienda Ospedaliera Universitaria di Ferrara
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided